CLINICAL TRIAL: NCT00318448
Title: Efficacy, Safety and Tolerability of Zolpidem in the Treatment of Children Aged 6 to 17 Years With ADHD-Associated Insomnia. A Multicentre, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Efficacy, Safety, and Tolerability of Ambien (Zolpidem) in the Treatment of Children Ages 6 to 17 With Attention Deficit Hyperactivity Disorder (ADHD)-Associated Insomnia
Acronym: Zolkids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6820
Record Dates: First submitted 2006-03-14; First posted 2006-04-26 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Child Psychology; Pediatric Psychology; Insomnia; Sleeplessness
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Zolpidem (SL800750)

SUMMARY:
There has been an increased interest in the association between ADHD and sleep disorders over the past years. A high incidence of sleep disturbance, ranging from 10% to 70%, has been identified in ADHD children regardless of whether or not they are receiving stimulant therapy. This study will assess the safety and efficacy of zolpidem in children with ADHD associated insomnia.

DETAILED DESCRIPTION:
The study is being conducted in the United States. It consists of 3 segments:

* Segment A: 2 to 21 day screening period
* Segment B: 8-week double-blind treatment period
* Segment C: 1-week follow-up period

Subjects will have a polysomnography in a sleep lab two times during the study (at baseline and between visit 4-5) and also be required to wear an actigraphy monitoring tool. There will be several questionnaires completed throughout the study: CGI-child, CGI-parent/legal guardian, ADHD Rating Scale-IV, and the Pediatric Daytime Sleepiness Scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 6 and 17 years, inclusive
* Children with diagnosed ADHD (as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision [DSM-IV-TR] criteria)
* Complaint of childhood insomnia as defined by repeated difficulty with sleep initiation or consolidation that occurs despite adequate age, appropriate time, and opportunity for sleep
* The sleep disturbance must not be attributable to either the direct physiologic effect of drug abuse or misuse of a prescribed medication.
* Subjects should be stabilized on all long-term therapy, including treatment of ADHD, for at least one month prior to study entry.
* Subjects, if females of childbearing potential (as determined by the initiation of menses), must have confirmed negative pregnancy test prior to randomization and be using a recognized effective method of birth control (oral, implant, depot or transdermal oestroprogestatives, intrauterine device, double-barrier with spermicide). Abstinence is an acceptable method of birth control for this study.

Exclusion Criteria:

* Mental retardation
* Autistic spectrum disorder
* A history of sleep apnea
* A history of bipolar disorder, conduct disorder, major depression, or generalized anxiety disorder (not obsessive compulsive disorder), as determined by clinical interview and DSM-IV-TR criteria
* Current history of substance abuse/dependence
* Known hypersensitivity to zolpidem or previous adverse experience with zolpidem
* Pregnant or breast-feeding
* Current use of hypnotics, antihistamines, melatonin, herbal products, or other sleep aids

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Latency to persistent sleep (LPS) measured by polysomnography

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) Severity and Global Improvement item scores (from child and parent/legal guardian scales)
Actigraphy measures of sleep characteristics
ADHD Rating Scale-IV
School tardiness/Attendance Reports
Adverse events
PE, lab

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Canada

REFERENCES:
- [Derived] Blumer JL, Findling RL, Shih WJ, Soubrane C, Reed MD. Controlled clinical trial of zolpidem for the treatment of insomnia associated with attention-deficit/ hyperactivity disorder in children 6 to 17 years of age. Pediatrics. 2009 May;123(5):e770-6. doi: 10.1542/peds.2008-2945. PMID 19403468